CLINICAL TRIAL: NCT04508634
Title: Comparison of the Clinical Efficacy of Laparoscopic Sleeve Gastrectomy and Metformin in the Treatment of Obese Patients With Polycystic Ovary Syndrome
Brief Title: Treating Obese PCOS Patients With LSG vs. Met
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Zhang Manna, Department of Endocrinology & Metabolism, Shanghai 10th People's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LSG vs. Met in PCOS
Record Dates: First submitted 2020-08-07; First posted 2020-08-11 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: laparoscopic sleeve gastrectomy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laparoscopic sleeve gastrectomy (Experimental): laparoscopic sleeve gastrectomy
  Interventions: Procedure: laparoscopic sleeve gastrectomy
- Metformin Group (Active Comparator): Metformin Group
  Interventions: Drug: Metformin Pill

INTERVENTIONS:
Procedure: laparoscopic sleeve gastrectomy — laparoscopic sleeve gastrectomy
  Other Names: Sleeve Operation
  Arms: laparoscopic sleeve gastrectomy
Drug: Metformin Pill — Metformin 1000mg bid
  Arms: Metformin Group

SUMMARY:
Polycystic ovary syndrome (PCOS) is a common endocrine disorder, with a prevalence of 5% to 15% in premenopausal women. Patients with PCOS presents as abnormal menstruation, ovulation disorders and/or hyperandrogenemia, and often accompanied by insulin resistance and other metabolic abnormalities. Sleeve gastrectomy was an effective threapy for severe obesity patients. This study will evaluate the clinical efficacy of sleeve gastrectomy for obese patients with PCOS. Mealwhile, the specific mechanism of sleeve gastrectomy for improving obese patients with PCOS will be explored through multi-group analysis.

ELIGIBILITY:
Inclusion Criteria:

* female aged 18- 45;
* meet Rotterdam criteria;
* BMI ≥ 28 kg /m2.

Exclusion Criteria:

* Women who are pregnant or have a pregnancy plan within six months;
* Women who are reluctant to undergo metabolic surgery;
* Congenital adrenocortical hyperplasia;
* Hyperprolactinemia;
* Hyperthyroidism or hypothyroidism;
* Abnormal liver function (≥ 3 times of the upper limit of normal range); abnormal · Rrenal function (GFR<60ml/min/1.73m2);
* Adrenal or ovarian tumors secreting androgens;
* Used contraceptives, metformin, GLP-1RA, pioglitazone and contraceptives in the last 3 month.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
HOMA-IR | 3 months
  Insulin resistance index
Screening of metabolites in plasma concentration in fasting condition | 3 months
  The investigators will perform metabolites to identify the changes that may give rise to the disease.
Screening of transcriptome profile in plasma concentration in fasting condition | 3 months
  The investigators will perform transcriptome profile to identify the changes that may give rise to the disease.
Screening of Microbiome in faeces | 3 months
  The investigators will perform Microbiome to identify the changes that may give rise to the disease.

SECONDARY OUTCOMES:
menstrual cycles | 3 months
  menstrual frequency
Gonadotropin level | 3 months
  LH(IU/L) , FSH (IU/L),
testosterone | 3 months
  total testosterone (nmol/L), testosterone (nmol/L)
SHBG level | 3 months
  SHBG (nmol/L).
FINS | 3 months
  fasting insulin (IU/L)
TC | 3 months
  Total cholesterol (mmol/L)
TG | 3 months
  Triglycerides (mmol/L)
HDL-c | 3 months
  high-density lipoprotein cholesterol (mmol/L)
LDL-c | 3 months
  low-density lipoprotein cholesterol (mmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Shen Qu, Dr, Study Chair — Shang hai Tenth People's Hospital
Locations (1):
- Shanghai Tenth People' Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No